CLINICAL TRIAL: NCT00255151
Title: A Phase 3 Study to Evaluate the Safety and Efficacy of Dexlansoprazole MR (60 mg QD and 90 mg QD) Compared to Placebo in Maintenance of Healing in Subjects With Healed Erosive Esophagitis
Brief Title: Comparison of Dexlansoprazole MR to Placebo on the Ability to Maintain Healing in Subjects With Healed Erosive Esophagitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: T-EE04-087; U1111-1114-1767 (Registry Identifier: WHO)
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Results first posted 2009-08-28 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Esophagitis, Reflux; Esophagitis, Peptic
Keywords: Erosive Esophagitis
MeSH Terms: conditions — Esophagitis, Peptic | interventions — Dexlansoprazole; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dexlansoprazole MR 60 mg QD (Experimental)
  Interventions: Drug: Dexlansoprazole MR
- Dexlansoprazole MR 90 mg QD (Experimental)
  Interventions: Drug: Dexlansoprazole MR
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexlansoprazole MR — Dexlansoprazole MR 60 mg, capsules, orally, once daily for up to six months.
  Other Names: TAK-390MR; Dexilant; Kapidex
  Arms: Dexlansoprazole MR 60 mg QD
Drug: Dexlansoprazole MR — Dexlansoprazole MR 90 mg, capsules, orally, once daily for up to six months.
  Other Names: TAK-390MR; Kapidex; Dexilant
  Arms: Dexlansoprazole MR 90 mg QD
Drug: Placebo — Dexlansoprazole placebo-matching capsules, orally, once daily for up to six months.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the ability of once-daily (QD) treatment with Dexlansoprazole modified-release (MR) 60 mg and 90 mg and placebo in maintaining healing of erosive esophagitis (EE).

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, multi-center, placebo-controlled, 6 month maintenance study. The study is designed to compare the efficacy and safety of daily Dexlansoprazole MR (60 mg and 90 mg) with that of placebo, in maintaining healing of erosive esophagitis.

Because the development plan for Dexlansoprazole MR formulation was revised, the results of 2 identical studies, T-EE04-086 (NCT00255164) and T-EE04-087 (this study, NCT00255151), were combined and analyzed as a single larger study referred to as study T-EE04-086. A total of 451 subjects were included in the combined analysis: 237 subjects were enrolled into Study T-EE04-086, and 214 subjects were enrolled into Study T-EE04-087.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have successfully completed the Phase 3 Study T-EE04-084 (NCT00251693) or T-EE04-085 (NCT00251719); and have healed esophageal erosions proven by endoscopy. Complete healing was assessed for change in LA Esophagitis Classification grades A, B, C, or D to healed (defined as anything less than the criterion for Grade A). The subject was counted as healed if endoscopy findings did not meet the Grade A criterion.

Exclusion Criteria:

* Use of prescription or nonprescription proton pump inhibitors (PPIs), histamine (H2) receptor antagonists, sucralfate, misoprostol, or prokinetics throughout the study
* Use of antacids (except for study supplied) throughout the study.
* Subjects using drugs with significant anticholinergic effects such as tricyclics who cannot stay on a stable dose throughout the study.
* Need for continuous anticoagulant therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2006-01; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Takeda
Locations (100):
- United States (100):
  - Anniston, Alabama
  - Hueytown, Alabama
  - Huntsville, Alabama
  - Tallassee, Alabama
  - Tuscaloosa, Alabama
  - Tucson, Arizona
  - Little Rock, Arkansas
  - North Little Rock, Arkansas
  - Azusa, California
  - Carmichael, California
  - Cypress, California
  - Fresno, California
  - Los Angeles, California
  - Modesto, California
  - Newport Beach, California
  - Oakland, California
  - Orange, California
  - San Diego, California
  - Santa Maria, California
  - Littleton, Colorado
  - Longmont, Colorado
  - Wheat Ridge, Colorado
  - Bristol, Connecticut
  - Newark, Delaware
  - Fort Myers, Florida
  - Miami, Florida
  - Naples, Florida
  - New Smyrna Beach, Florida
  - Ocala, Florida
  - Pembroke Pines, Florida
  - Port Orange, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Zephyrhills, Florida
  - Atlanta, Georgia
  - Champaign, Illinois
  - Moline, Illinois
  - North Chicago, Illinois
  - Oak Forest, Illinois
  - Springfield, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Newburgh, Indiana
  - Davenport, Iowa
  - Kansas City, Kansas
  - Wichita, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Chevy Chase, Maryland
  - Prince Frederick, Maryland
  - Jackson, Mississippi
  - Jefferson City, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Missoula, Montana
  - Egg Harbor, New Jersey
  - Albuquerque, New Mexico
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - High Point, North Carolina
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Bismarck, North Dakota
  - Akron, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Mogadore, Ohio
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Warwick, Rhode Island
  - Anderson, South Carolina
  - Mt. Pleasant, South Carolina
  - Sioux Falls, South Dakota
  - Chattanooga, Tennessee
  - Germantown, Tennessee
  - Jackson, Tennessee
  - Johnson City, Tennessee
  - Kingsport, Tennessee
  - Amarillo, Texas
  - Conroe, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Odessa, Texas
  - Pharr, Texas
  - Seguin, Texas
  - Temple, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Bellevue, Washington
  - Lakewood, Washington
  - Tacoma, Washington
  - Milwaukee, Wisconsin

REFERENCES:
- [Result] Howden CW, Larsen LM, Perez MC, Palmer R, Atkinson SN. Clinical trial: efficacy and safety of dexlansoprazole MR 60 and 90 mg in healed erosive oesophagitis - maintenance of healing and symptom relief. Aliment Pharmacol Ther. 2009 Nov 1;30(9):895-907. doi: 10.1111/j.1365-2036.2009.04119.x. Epub 2009 Aug 14. PMID 19681809
- See also: For the Dexilant package insert refer to this link — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=9efb34b3-fb69-4190-a2be-a90b8cb94e25&filetypecode=DEXILANTPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 105 sites in the United States; date of first dose (04 January 2006; date of last procedure: 14 November 2006).
Pre-assignment Details: Subjects had to have endoscopically proven healed erosive esophagitis (EE) after 4 to 8 weeks of treatment with lansoprazole 30 mg once-daily (QD), dexlansoprazole modified release (MR) 60 mg QD, or dexlansoprazole MR 90 mg QD in the EE healing studies, T-EE04-084 (NCT00251693) and T-EE04-085 (NCT00251719).
Groups:
- Placebo QD: Placebo capsules, orally, once daily for up to 6 months.
- Dexlansoprazole MR 60 mg QD: Dexlansoprazole MR 60 mg, capsules, orally, once daily for up to 6 months.
- Dexlansoprazole MR 90 mg QD: Dexlansoprazole MR 90 mg, capsules, orally, once daily for up to 6 months.
Period: Overall Study
Arm/Group | Placebo QD | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Started | 140 | 159 | 152
Completed | 17 | 110 | 103
Not Completed | 123 | 49 | 49
Not completed — Adverse Event | 10 | 6 | 9
Not completed — Lost to Follow-up | 4 | 3 | 4
Not completed — Withdrawal by Subject | 18 | 17 | 8
Not completed — Noncompliance | 0 | 1 | 2
Not completed — Subject Request/Subject Unavailable | 1 | 1 | 2
Not completed — Relapse of Erosive Esophagitis | 78 | 16 | 12
Not completed — Possible Barrett's Esophagus | 1 | 3 | 8
Not completed — Esophageal Stricture | 0 | 0 | 1
Not completed — Therapeutic Failure | 11 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo QD | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD | Total
Number analyzed (Participants) | 140 | 159 | 152 | 451
Age Continuous [Mean (Standard Deviation); unit: years] | 48.2 (12.88) | 49.7 (12.66) | 48.8 (13.76) | 48.9 (13.09)
Age, Customized [Number; unit: participants]
  <45 years | 48 | 55 | 56 | 159
  45 to <65 years | 81 | 86 | 81 | 248
  ≥65 years | 11 | 18 | 15 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 76 | 70 | 216
  Male | 70 | 83 | 82 | 235
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 1 | 5
  Asian | 2 | 3 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 17 | 11 | 39
  White | 124 | 135 | 136 | 395
  More than one race | 1 | 2 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 19 | 14 | 48
  Not Hispanic or Latino | 125 | 140 | 138 | 403
  Unknown or Not Reported | 0 | 0 | 0 | 0
Baseline Los Angeles (LA) Classification Grade for Erosive Esophagitis (EE) [Number; unit: participants] — Baseline values from Studies T-EE04-084 (NCT00251693)and T-EE04-085 (NCT00251719), with severity of EE increasing from Grade A to Grade D.
  participants
    A: ≥1 mucosal break <5 mm | 58 | 60 | 54 | 172
    B: ≥1 mucosal break ≥5 mm | 48 | 61 | 58 | 167
    C: ≥1 mucosal break <75% of circumference | 28 | 33 | 32 | 93
    D: ≥1 mucosal break ≥75% of circumference | 6 | 5 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Maintained Complete Healing of Erosive Esophagitis as Assessed by Endoscopy - Crude Rate Analysis.
Description: Crude rates analyzed maintenance of healed EE from baseline of this study and considered prematurely discontinued subjects as relapsed.
Time Frame: 6 months
Population: The crude rate analysis was performed on intent-to-treat (ITT) subjects (subjects from Studies T-EE04-084 or T-EE04-085 with endoscopically proven healed EE who received at least 1 dose of study drug in this study and did not have a gap of >7 days between the EE healing studies and this study) with at least one endoscopy in this maintenance study.
Measure: Number; unit: Percentage of Subjects
Arm/Group | Placebo QD | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 112 | 152 | 138
Percentage of Subjects | 14.3 [8.4 to 22.2] | 66.4 [58.3 to 73.9] | 64.5 [55.9 to 72.4]
Statistical Analysis 1: Comparison: Placebo QD vs Dexlansoprazole MR 60 mg QD; Test type: Superiority or Other; p < 0.00001, Fisher Exact — Hochberg's method was used to ensure that the overall 0.0025 level of significance was maintained for the pairwise comparisons between each dexlansoprazole MR dose and placebo
Statistical Analysis 2: Comparison: Placebo QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p < 0.00001, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.80473, Fisher Exact — Statistical significance was determined at 0.0025 level without adjustment for multiple comparisons

2. Secondary Outcome: Percentage of Days Without Daytime or Nighttime Heartburn as Assessed by Daily Diary-Median.
Description: The percentage was calculated as the days that were heartburn-free out of the total number of days for which either a daytime or nighttime result was reported.
Time Frame: 6 months
Population: The analysis of 24-hour heartburn-free days was performed on ITT subjects with at least one daytime or nighttime heartburn Yes/No question answered during treatment.
Measure: Median (Inter-Quartile Range); unit: Percentage of Days
Arm/Group | Placebo QD | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 133 | 157 | 147
Percentage of Days | 19.2 (29.3) [5.0 to 52.0] | 95.8 (30.7) [76.9 to 99.1] | 94.4 (30.0) [67.1 to 99.4]
Statistical Analysis 1: Comparison: Placebo QD vs Dexlansoprazole MR 60 mg QD; Test type: Superiority or Other; p < 0.00001, Wilcoxon (Mann-Whitney) — The 0.0025 level of significance for this secondary endpoint was controlled using Hochberg's method for comparisons of each dexlansoprazole MR dose to placebo
Statistical Analysis 2: Comparison: Placebo QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p < 0.00001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.76046, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.0025 level without adjustment for multiple comparisons

3. Secondary Outcome: Percentage of Days Without Daytime or Nighttime Heartburn as Assessed by Daily Diary-Mean.
Description: The percentage was calculated as the days that were heartburn-free out of the total number of days for which either a daytime or nighttime result was marked
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of Days
Arm/Group | Placebo QD | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 133 | 157 | 147
Percentage of Days | 29.5 (29.3) | 79.7 (30.7) | 79.2 (30.0)

4. Primary Outcome: Percentage of Subjects Who Maintained Complete Healing of Erosive Esophagitis as Assessed by Endoscopy - Life Table Method
Description: Percentage of subjects who maintained complete healing of erosive esophagitis as assessed by endoscopy. In the life table method, subjects without post-baseline endoscopy were included as censored; subjects who did not have a recurrence of EE and did not complete the study were also considered censored.
Time Frame: 6 months
Population: Life table method for the maintenance rate of healed EE was performed on ITT subjects and included subjects without post-baseline endoscopy as censored.
Measure: Number; unit: Percentage of Subjects
Arm/Group | Placebo QD | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 140 | 159 | 152
Percentage of Subjects | 25.7 | 86.6 | 82.1
Statistical Analysis 1: Comparison: Placebo QD vs Dexlansoprazole MR 60 mg QD; Test type: Superiority or Other; p < 0.00001, Log Rank — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p < 0.00001, Log Rank — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.37161, Log Rank — Statistical significance was determined at 0.0025 level without adjustment for multiple comparisons

5. Secondary Outcome: Percentage of Days Without Nighttime Heartburn as Assessed by Daily Diary-Median.
Description: The percentage was calculated as the nights that were heartburn-free out of the total number of days for which a nighttime result was marked.
Time Frame: 6 months
Population: The analysis was performed on ITT subjects with at least one nighttime heartburn Yes/No question answered during treatment.
Measure: Median (Inter-Quartile Range); unit: Percentage of Days
Arm/Group | Placebo QD | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 133 | 157 | 147
Percentage of Days | 50.0 (35.3) [14.8 to 81.3] | 98.3 (25.5) [90.6 to 100.0] | 97.1 (26.3) [83.3 to 100.0]
Statistical Analysis 1: Comparison: Placebo QD vs Dexlansoprazole MR 60 mg QD; Test type: Superiority or Other; p < 0.00001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p < 0.00001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.59700, Wilcoxon (Mann-Whitney) — Statistical significance was determined at the 0.0025 level without adjustment for multiple comparisons

6. Secondary Outcome: Percentage of Days Without Nighttime Heartburn as Assessed by Daily Diary-Mean.
Description: as for outcome 5
Time Frame: 6 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of Days
Arm/Group | Placebo QD | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 133 | 157 | 147
Percentage of Days | 48.3 (35.3) | 87.1 (25.5) | 85.4 (26.3)

ADVERSE EVENTS:
Arm/Group | Placebo QD | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Serious Adverse Events (participants affected / at risk) | 0 | 2 | 5
Other Adverse Events (participants affected / at risk) | 7 | 33 | 25
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Placebo QD | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Coronary Artery Disorders Not Elsewhere Classified (NEC) (Cardiac disorders) | 0/140 | 0/159 | 1/152
Acute and Chronic Pancreatitis (Gastrointestinal disorders) | 0/140 | 0/159 | 1/152
Pain and Discomfort NEC (General disorders) | 0/140 | 1/159 | 0/152
Non-site Specific Injuries NEC (Injury, poisoning and procedural complications) | 0/140 | 0/159 | 1/152
Musculoskeletal and Connective Tissue Signs and Symptoms NEC (Musculoskeletal and connective tissue disorders) | 0/140 | 0/159 | 1/152
Breast and Nipple Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/140 | 0/159 | 1/152
Uterine Disorders NEC (Reproductive system and breast disorders) | 0/140 | 1/159 | 0/152
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Placebo QD | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Diarrhoea (Excluding [Excl] Infective) (Gastrointestinal disorders) | 1/140 | 10/159 | 10/152
Flatulence, Bloating and Distension (Gastrointestinal disorders) | 0/140 | 8/159 | 3/152
Gastritis (Excl Infective) (Gastrointestinal disorders) | 1/140 | 10/159 | 6/152
Gastrointestinal and Abdominal Pains (Excl Oral and Throat) (Gastrointestinal disorders) | 2/140 | 10/159 | 6/152
Upper Respiratory Tract Infections (Infections and infestations) | 5/140 | 4/159 | 7/152

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.